CLINICAL TRIAL: NCT04041830
Title: Validation of a French-version of the Leeds Food Preference Questionnaire in Normal Weight and Patients With Obesity
Acronym: LFPQ-F
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sanitary conditions and material restrictions imposed by the CHU and by the university laboratories drastically hampered the realization of this work (with restricted access to the laboratory/department).
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Appetite Control and Energy Balance Research Group, UNiversity of Leeds, Leeds, UK (Unknown); Laboratoire AME2P. Campus universitaire des cezeaux, 63170 Aubiere, Cedex (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2019 GENTES; 2019-A00853-54 (Other: 2019-A00853-54)
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Normal Weight Adults; Adults With Obesity
Keywords: Appetite; Food Reward; Methodological approach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NW (Normal Weight) (Experimental): 20 to 55 years old lean adults
  Interventions: Behavioral: Visit 1; Behavioral: Visit 2
- OBESE (Experimental): 20 to 55 years old adults with obesity
  Interventions: Behavioral: Visit 1; Behavioral: Visit 2

INTERVENTIONS:
Behavioral: Visit 1 — the participants will fill in the LFPQ questionnaire before and after a lunch test meal
Behavioral: Visit 2 — this is a replication of Visit 1, testing the reproducibility of the LFPQ and of its response to a meal.

SUMMARY:
While Food reward is an important component of the appetite control to consider, there is actually no tool that has been developed in French to perform its evaluation.

The Leeds Food Preference Questionnaire (LFPQ) is a validated and recognized tool to assess food reward, being however developed for British populations.

The aim of this work is to validate a French version of the LFPQ among lean and obese adults.

DETAILED DESCRIPTION:
50 lean and 50 patients with obesity between 20 and 55 years old (50% women and 50% men), will be recruited. After an evaluation of their body composition by impedance meter, and of their dietary status by questionnaires (TFEQ/DEBQ), they will be asked to perform twice the same experimental sessions. They will be asked during this session to arrive at 08:00 am after a 12-hour fast and will receive a calibrated breakfast. Before and after a lunch calibrated meal, they will be asked to perform the French version of the computerized questionnaire LFPQ. Appetite feelings will be assessed at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30 and 38 kg.m² for the obese patients and 20 and 25 for the lean ones.
* registered to the national social security system
* Signed consent

Exclusion Criteria:

* eating disorders
* metabolic disease such as hypertension and Type 2 diabetes

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2019-12-08 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Change in Food reward | day 1 , day 8
  The participants will be asked to complete the developed French version of the computer-based procedure to measure food reward (Leeds Food Preference Questionnaire; LFPQ) (Finlayson, King et al. 2008).

SECONDARY OUTCOMES:
Body fat mass | day 0
  the percentage of body fat and the quantity of fat mass will be assessed using Bio-impedance (BIA)
Body fat and fat free mass | day 0
  the percentage of body fat free and the quantity of fat free mass will be assessed using Bio-impedance (BIA)
Dietary status | day 0
  the level of dietary restriction/disinhibition will be assessed using the TFEQ questionnaire.
Dietary status | day 0
  the level of dietary restriction/disinhibition will be assessed using the DEBQ questionnaire.
Hunger | day 1, day 1 + 30minutes, day 1+60minutes, day 1+ 90minutes , day 8, day 8 + 30minutes, day 8+60minutes, day 8+ 90minutes
  the hunger sensation will be assessed using visual analogue scales of 150 mm.
Satiety | dday 1, day 1 + 30minutes, day 1+60minutes, day 1+ 90minutes , day 8, day 8 + 30minutes, day 8+60minutes, day 8+ 90minutes
  the Satiety sensation will be assessed using visual analogue scales of 150 mm.
desire to eat | day 1, day 1 + 30minutes, day 1+60minutes, day 1+ 90minutes , day 8, day 8 + 30minutes, day 8+60minutes, day 8+ 90minutes
  the desire to eat sensation will be assessed using visual analogue scales of 150 mm.
Prospective Food consumption | day 1, day 1 + 30minutes, day 1+60minutes, day 1+ 90minutes , day 8, day 8 + 30minutes, day 8+60minutes, day 8+ 90minutes
  the Prospective Food consumption sensation will be assessed using visual analogue scales of 150 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Elodie Gentes, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France